CLINICAL TRIAL: NCT03530228
Title: A Randomized, Open-label, Active-controlled, Single/Multiple-dose Phase 1 Clinical Trial to Evaluate Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of Tegoprazan After Oral Administration in Healthy Male Subjects
Brief Title: A Phase 1 Study of Tegoprazan on Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_APA_109
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pharmacodynamics; Pharmacokinetics; Healthy Male Volunteers
MeSH Terms: interventions — tegoprazan; Esomeprazole

STUDY DESIGN:
Intervention Model Description: Cohort 1: crossover Cohort 2: parallel Cohort 3: single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Treatment A: Tegoprazan (C1) (Experimental): Tegoprazan QD, oral administration
  Interventions: Drug: Tegoprazan (C1)
- Treatment B: Tegoprazan (C1) (Experimental): Tegoprazan QD, oral administration
  Interventions: Drug: Tegoprazan (C1)
- Treatment C: Tegoprazan (C1) (Experimental): Tegoprazan BID, oral administration
  Interventions: Drug: Treatment C: Tegoprazan (C1)
- Group 1: Tegoprazan (C2) (Experimental): Tegoprazan QD, oral administration, for 7 days
  Interventions: Drug: Tegoprazan (C2)
- Group 2: Tegoprazan (C2) (Experimental): Tegoprazan QD, oral administration, for 7 days
  Interventions: Drug: Tegoprazan (C2)
- Group 3: Esomeprazole (C2) (Active Comparator): Esomeprazole QD, oral administration, for 7 days
  Interventions: Drug: Esomeprazole (C2)
- Tegoprazan (C3) (Experimental): Tegoprazan QD, oral administration
  Interventions: Drug: Tegoprazan (C3)

INTERVENTIONS:
Drug: Tegoprazan (C1) — Tegoprazan QD, oral administration. Treatment A
  Arms: Treatment A: Tegoprazan (C1)
Drug: Tegoprazan (C1) — Tegoprazan QD, oral administration. Treatment B
  Arms: Treatment B: Tegoprazan (C1)
Drug: Treatment C: Tegoprazan (C1) — Tegoprazan BID, oral administration
  Arms: Treatment C: Tegoprazan (C1)
Drug: Tegoprazan (C2) — Tegoprazan QD, oral administration, for 7 days. Group 1
  Arms: Group 1: Tegoprazan (C2)
Drug: Tegoprazan (C2) — Tegoprazan QD, oral administration, for 7 days. Group 2
  Arms: Group 2: Tegoprazan (C2)
Drug: Esomeprazole (C2) — Esomeprazole QD, oral administration, for 7 days. Group 3
  Arms: Group 3: Esomeprazole (C2)
Drug: Tegoprazan (C3) — Tegoprazan QD, oral administration
  Arms: Tegoprazan (C3)

SUMMARY:
A randomized, open-label, active-controlled, single/multiple-dose phase 1 clinical trial to evaluate pharmacokinetics/pharmacodynamics and safety/tolerability of tegoprazan after oral administration in healthy male subjects

DETAILED DESCRIPTION:
* To evaluate the pharmacokinetics and pharmacodynamics of single oral dose of tegoprazan between dose groups in healthy H. pylori negative males.
* To evaluate the pharmacokinetics and pharmacodynamics of multiple oral dose of tegoprazan under the fed state in healthy H. pylori negative males.
* To evaluate the pharmacokinetics and pharmacodynamics of single oral dose of tegoprazan in healthy H. pylori positive males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged ≥ 19 years and ≤ 50 years
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2 at the time of screening

Exclusion Criteria:

* Presence or history of clinically significant diseases
* Presence or history of gastrointestinal disorder (gastric ulcer, GERD, - Crohn's disease, etc.)
* Hypersensitivity to drugs containing study drug or proton pump inhibitor and other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity
* Serologic test positive
* Abnormal obstacle to insertion and maintenance of pH meter catheter
* History of drug abuse
* Excessive caffeine intake or persistent alcohol intake
* Not use of a medically acceptable method of contraception

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
AUC(0-24h) of tegoprazan | up to 7 days
  Area Under the Curve(0-24h) of tegoprazan
Cmax of tegoprazan | up to 7 days
  Maximum Plasma Concentration of tegoprazan
Gastric pH | up to 7 days
  Gastric pH
Serum gastrin concentration | up to 7 days
  Serum gastrin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea